CLINICAL TRIAL: NCT05809557
Title: Effect of an EMR Chemotoxicity Risk Calculator Availability To Decrease Chemotherapy Toxicity in Adults With Cancer
Brief Title: EMR Chemotoxicity Risk Calculator To Decrease Chemotherapy Toxicity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2022LS125; STUDY00015357 (Other: IRB)
Record Dates: First submitted 2023-03-30; First posted 2023-04-12 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Oncology; Chemotherapeutic Toxicity; Metastatic Solid Tumor
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Intervention Model Description: Providers, who were selected based on having at least 20 new patients with metastatic solid tumors in a 6-month period in 2021, will be randomized in a 1:1 ratio, stratified by quartiles of patient volume.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (Placebo Comparator)
  Interventions: Other: Oncology Consultation
- Chemotherapy Toxicity Tool (Experimental)
  Interventions: Other: Chemotherapy toxicity tool; Other: Oncology Consultation

INTERVENTIONS:
Other: Chemotherapy toxicity tool — CARG is an EMR based tool that informs medical oncologists visiting a patient for the first time of potential risk of chemotherapy toxicity. This intervention will make available a simple calculator which includes: Gender, Height and weight, Cancer Subtype, Hemoglobin, How is your hearing (with hearing aid, if needed)?, Number of falls in the past 6 months, Can you take your own medicines, Does your health limit you in walking one block., During the past 4 weeks, how much of the time has your physical health or emotional problems interfered with your social activities (like visiting with friends, relatives, etc.)? and Glomerular filtration rate.
  The CARG chemotoxicity calculator will be built into the patient navigator and its use will be assessed on a monthly basis and used to inform iteration.
  Other Names: CARG
  Arms: Chemotherapy Toxicity Tool
Other: Oncology Consultation — Oncologists will consult new patient with a new diagnosis of cancer.

SUMMARY:
This study will formally test the quality improvement intervention of an EMR based tool that informs medical oncologists visiting a patient for the first time of potential risk of chemotherapy toxicity.

ELIGIBILITY:
Inclusion Criteria:

* New outpatient visits with a medical oncologist following a new diagnosis of cancer and no prior history of chemotherapy treatment.
* aged > 65 will be included.

Exclusion Criteria:

* Patients who opt out of clinical research will be excluded from analysis, but not the intervention (which will be applied to all patients). Specifically, as sometimes opt-in/opt out status is coded ambiguously in the data we will only analyze results of patients with clear opt in and no history of opt out.
* Patients with no EHR data after initial oncologist appointment.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 34 (Actual)
Dates: Start 2023-01-09 (Actual); Primary Completion 2023-06-09 (Actual); Study Completion 2024-01-09 (Actual)

PRIMARY OUTCOMES:
Unplanned hospitalization rate | Within 3 months of the Index Visit with the oncologist
  Measured at the patient level as a binary outcome (yes/no) based on date of initial visit with the oncologist.

SECONDARY OUTCOMES:
Healthcare contact days | Within 3 and 6 months of the Index Visit with the oncologist
  Measured at the patient level as a continuous outcome (number of days).
Chemotherapy use rate | Within 3 months of the Index Visit with the oncologist
  Measured at the patient level as a binary outcome (yes/no) if patient ever received systemic cancer-directed treatment.
Chemotherapy modification rate | Within 3 months of the Index Visit with the oncologist
  Measured at the patient level as a binary outcome (yes/no) if patient had dose, schedule, or number of chemotherapy changed.
Palliative Care Referral | Within 6 months of the Index Visit with the oncologist
  Measured at the patient level as a binary outcome (yes/no) based on presence of a scheduled palliative care appointment
Chemotherapy toxicity tool use rate | Within 3 months of the Index Visit with the oncologist
  Measured at the patient level as a binary outcome (yes/no) based on whether the oncologist used the tool for that patient.

CONTACTS AND LOCATIONS:
Locations (1):
- Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
All data will be housed as subset within the existing Center for Learning Health System Science/Center for Quality Outcomes, Discovery and Evaluation database covered by IRB 597 Protocol: STUDY00014481. Patient level data will not be shared with anyone outside the study team. Aggregated data will be shared with quality officials, hospital administrators, and more broadly disseminated in academic meetings and for publication.